CLINICAL TRIAL: NCT05731024
Title: Protocol for Comparing Closed-loop syncHronization vErsuS convenTional Synchronization In sPontaneously Breathing Pediatric Patients (CHESTSIPP) - a Randomized Cross-over Study
Brief Title: Closed-loop Synchronization Versus Conventional Synchronization
Acronym: CHESTSIPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Hasan ağın, Professor, Dr. Behcet Uz Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02019336
Record Dates: First submitted 2023-02-03; First posted 2023-02-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Failure; Pediatric Respiratory Distress Syndrome
Keywords: Acute respiratory failure (ARF); Pediatric acute respiratory distress syndrome (PARDS); Closed-loop; synchronization; patient ventilator asynchrony
MeSH Terms: conditions — Respiratory Distress Syndrome; Patient-Ventilator Asynchrony

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Close-loop synchronization controller (Experimental): One-hour period where the pressure support of spontaneous effort will be automatically titrated based on pressure and flow waveform analysis obtained from the patient during SPONT mode.
  Interventions: Device: close-loop synchronization controller with SPONT mode
- Conventional (Active Comparator): One-hour period where the synchronization of pressure support of patient effort during SPONT mode will be manually set.
  Interventions: Device: Conventional synchronization settings with SPONT mode

INTERVENTIONS:
Device: close-loop synchronization controller with SPONT mode — One-hour period where the pressure support of spontaneous breath will be automatically titrated based on pressure and flow waveform analysis obtained from the patient.
  Arms: Close-loop synchronization controller
Device: Conventional synchronization settings with SPONT mode — One-hour period where the pressure support of spontaneous breath will be manually set.
  Arms: Conventional

SUMMARY:
A prior research indicated that asynchrony between the patient and ventilator occurred in 33 percent of 19,175 breaths, and was seen in every patient. The most prevalent kind of asynchrony was ineffective triggering (68%), followed by delayed termination (19%), double triggering (4%) and premature termination (3%). Asynchrony between the patient and ventilator increased considerably with decreasing levels of peak inspiratory pressure, positive end-expiratory pressure, and set frequency.Despite this, more asynchrony categories exist, and there is no widely accepted categorization. Major asynchronies, however, include auto trigger, ineffective effort, and double trigger, while minor asynchronies include early/late cycle, trigger delay, and spontaneous breaths during a mandatory breath. This study aims to compare the safety and efficacy of a closed-loop synchronization controller with conventional control of synchronization during invasive mechanical ventilation of spontaneous breathing of pediatric patients in a pediatric intensive care unit (PICU).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients older than 1 month and younger than18 years of age
* Hospitalized at the PICU with the intention of treatment with mechanical ventilation at least for the upcoming 3 hours with spontaneous breathing activity
* Written informed consent signed and dated by the patient or one relative in case that the patient is unable to consent, after full explanation of the study by the investigator and prior to study participation

Exclusion Criteria:

* Formalized ethical decision to withhold or withdraw life support
* Patient included in another interventional research study under consent
* Patient already enrolled in the present study in a previous episode of respiratory failure
* Pregnant woman
* Patients deemed at high risk for the need of transportation from PICU to another ward, diagnostic unit or any other hospital
* Hemodynamic instability defined as a need of continuous infusion of epinephrine or norepinephrine > 1 mg/h
* Not being able to obtain reference waveform

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Asynchrony Index | 1 hour
  [(major asynchronies+minor asynchronies )/(total number of breaths + ineffective efforts)]x100

SECONDARY OUTCOMES:
Major asynchronies | 1 hour
  [(major asynchronies)/(total number of breaths + ineffective efforts)]x100
Minor asynchronies | 1 hour
  [(minor asynchronies)/(total number of breaths + ineffective efforts)]x100
Comfort Behavioral Score | 1 hour
  The Comfort Behavioral Scale yields points based on scores obtained from the Comfort B Scale. Scores below 10 indicate that the patient may be over-sedated, while scores between 12 and 17 suggest that the patient is adequately comfortable. Scores above 17 may suggest that the patient is experiencing inadequate sedation
Leak | 1 hour
  Percentage of leak around endotrachel tube (%)
Mean SpO2 | 1 hour
  Mean peripheral oxygen saturation (%)
Mean EtCO2 | 1 hour
  Mean end-tidal carbon dioxide (mm Hg)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Agin, Professor, Principal Investigator — Behcet Uz Children's Hospital
Locations (4):
- Turkey (Türkiye) (4):
  - Aydin Obstetric and pediatrics Hospital, Aydin
  - Erzurum Regional Research and Training Hospital, Erzurum
  - Cam Sakura Research and Training Hospital, Istanbul
  - The Health Sciences University Izmir Behçet Uz Child Health and Diseases Research and Training Hospital, Izmir

REFERENCES:
- [Background] van Dijk J, Blokpoel RGT, Abu-Sultaneh S, Newth CJL, Khemani RG, Kneyber MCJ. Clinical Challenges in Pediatric Ventilation Liberation: A Meta-Narrative Review. Pediatr Crit Care Med. 2022 Dec 1;23(12):999-1008. doi: 10.1097/PCC.0000000000003025. Epub 2022 Jul 14. PMID 35830707
- [Background] Emeriaud G, Newth CJ; Pediatric Acute Lung Injury Consensus Conference Group. Monitoring of children with pediatric acute respiratory distress syndrome: proceedings from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5 Suppl 1):S86-101. doi: 10.1097/PCC.0000000000000436. PMID 26035368
- [Background] Blokpoel RG, Burgerhof JG, Markhorst DG, Kneyber MC. Patient-Ventilator Asynchrony During Assisted Ventilation in Children. Pediatr Crit Care Med. 2016 May;17(5):e204-11. doi: 10.1097/PCC.0000000000000669. PMID 26914624
- [Background] Colleti J Jr, Brunow de Carvalho W. Patient-Ventilator Asynchrony During Assisted Ventilation in Children: The Time to Rethink Our Knowledge. Pediatr Crit Care Med. 2016 Aug;17(8):811. doi: 10.1097/PCC.0000000000000793. No abstract available. PMID 27500623
- [Background] Vignaux L, Grazioli S, Piquilloud L, Bochaton N, Karam O, Jaecklin T, Levy-Jamet Y, Tourneux P, Jolliet P, Rimensberger PC. Optimizing patient-ventilator synchrony during invasive ventilator assist in children and infants remains a difficult task*. Pediatr Crit Care Med. 2013 Sep;14(7):e316-25. doi: 10.1097/PCC.0b013e31828a8606. PMID 23842584
- [Background] Blokpoel RGT, Burgerhof JGM, Markhorst DG, Kneyber MCJ. Trends in Pediatric Patient-Ventilator Asynchrony During Invasive Mechanical Ventilation. Pediatr Crit Care Med. 2021 Nov 1;22(11):993-997. doi: 10.1097/PCC.0000000000002788. PMID 34054119